CLINICAL TRIAL: NCT02319954
Title: Intra-operative Nasal Compression After Lateral Osteotomy to Minimize Post-operative Peri-orbital Ecchymosis and Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: HSREB 105768
Record Dates: First submitted 2014-12-14; First posted 2014-12-18 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Rhinoplasty; Ecchymosis
MeSH Terms: conditions — Ecchymosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compression (Active Comparator): Each patient will be randomized to receive compression of their nose on either the left or right for 5 continuous minutes after performing a lateral rhinotomy.
  Interventions: Procedure: Direct compression
- No compression (No Intervention): Each patient will serve as their own control with the other side not receiving any compression after a lateral rhinotomy.

INTERVENTIONS:
Procedure: Direct compression — Direct compression by the surgeon with their hands on the nasal sidewall
  Arms: Compression

SUMMARY:
Periorbital edema and ecchymosis are common morbidities in the post-operative period after rhinoplasty. Lateral osteotomy techniques used to reshape the bony nasal pyramid are large contributing factors to the degree of bruising and edema. This is due to injury to the angular vessels that are crossing the osteotomy sites. Depending on the degree of swelling and bruising, it can cause difficulty with visual acuity in the early post-operative period. Most importantly, this can be quite distressing to the patient and impact the time required to return to normal social activities. Numerous studies have examined various interventions to reduce periorbital swelling and ecchymosis. These include peri-operative steroids, lidocaine with epinephrine injections, fibrin sealant, permissive intra-operative hypotension and subperiosteal osteotomy techniques. Peri-operative steroids have been most extensively studied. Recent meta-analysis by Hatef et al, found that pre-operative steroids were effective for decreasing post-operative edema and ecchymosis. Steroids however, carry with it the risks of psychosis, immunosuppression, weight gain, uncontrolled blood glucose and avascular necrosis of the hip. As such, broadly applicable and cost-effective techniques to minimize post-operative edema and ecchymosis without the risk profile of steroids would be ideal. Taskin et al. recently examined the efficacy of the combination of intraoperative cold saline-soaked gauze compression and corticosteroids on rhinoplasty morbidity. The study group received compression with a cold saline soaked gauze to the nasal dorsum during the surgery and the control group received compression with a dry gauze. Both groups received a pre-operative dose of intravenous steroids. The study group had significantly less periorbital edema and ecchymosis on post-operative days 1, 3, 5 and 7. This study unfortunately did not examine the role of compression alone and the study was performed in the presence of steroids, which is not routinely utilized by all surgeons. As such, the proposed study will provide evidence for the use of direct compression intra-operatively after lateral osteotomy in order to reduce post-operative edema and ecchymosis. The findings of this study may provide a simple, effective and non-costly technique to minimize the morbidity of rhinoplasty.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (18 years old and greater) undergoing rhinoplasty requiring lateral osteotomy

Exclusion Criteria:

* Patients taking anti-coagulation medication, history of bleeding disorder and those who do not complete the follow-up schedule will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Periorbital edema and ecchymosis | up to 4 weeks
  The primary outcome of this study is periorbital edema and ecchymosis. Post-operative photographs will be graded by two staff Otolaryngologists and two senior Otolaryngology residents. Each evaluator will be presented a photograph of a patient and be asked to grade the degree of periorbital edema and ecchymosis for the left and right side. Previously published grading scales will be used. The evaluators will be blinded to the allocated side of nasal pressure and to the post-operative day of the photographs.

REFERENCES:
- [Background] Taskin U, Yigit O, Bilici S, Kuvat SV, Sisman AS, Celebi S. Efficacy of the combination of intraoperative cold saline-soaked gauze compression and corticosteroids on rhinoplasty morbidity. Otolaryngol Head Neck Surg. 2011 May;144(5):698-702. doi: 10.1177/0194599811400377. PMID 21493314
- [Background] Tuncel U, Turan A, Bayraktar MA, Erkorkmaz U, Kostakoglu N. Efficacy of dexamethasone with controlled hypotension on intraoperative bleeding, postoperative oedema and ecchymosis in rhinoplasty. J Craniomaxillofac Surg. 2013 Mar;41(2):124-8. doi: 10.1016/j.jcms.2012.06.003. Epub 2012 Jul 12. PMID 22795164
- [Background] Totonchi A, Guyuron B. A randomized, controlled comparison between arnica and steroids in the management of postrhinoplasty ecchymosis and edema. Plast Reconstr Surg. 2007 Jul;120(1):271-274. doi: 10.1097/01.prs.0000264397.80585.bd. PMID 17572575
- [Background] Hatef DA, Ellsworth WA, Allen JN, Bullocks JM, Hollier LH Jr, Stal S. Perioperative steroids for minimizing edema and ecchymosis after rhinoplasty: a meta-analysis. Aesthet Surg J. 2011 Aug;31(6):648-57. doi: 10.1177/1090820X11416110. PMID 21813878
- [Background] Gun R, Yorgancilar E, Yildirim M, Bakir S, Topcu I, Akkus Z. Effects of lidocaine and adrenaline combination on postoperative edema and ecchymosis in rhinoplasty. Int J Oral Maxillofac Surg. 2011 Jul;40(7):722-9. doi: 10.1016/j.ijom.2011.02.022. Epub 2011 Apr 1. PMID 21458231
- [Background] Kosucu M, Omur S, Besir A, Uraloglu M, Topbas M, Livaoglu M. Effects of perioperative remifentanil with controlled hypotension on intraoperative bleeding and postoperative edema and ecchymosis in open rhinoplasty. J Craniofac Surg. 2014 Mar;25(2):471-5. doi: 10.1097/SCS.0000000000000603. PMID 24531244
- [Background] Al-Arfaj A, Al-Qattan M, Al-Harethy S, Al-Zahrani K. Effect of periosteum elevation on periorbital ecchymosis in rhinoplasty. J Plast Reconstr Aesthet Surg. 2009 Nov;62(11):e538-9. doi: 10.1016/j.bjps.2008.05.047. Epub 2008 Oct 5. No abstract available. PMID 18838319
- [Background] Kara CO, Kara IG, Topuz B. Does creating a subperiosteal tunnel influence the periorbital edema and ecchymosis in rhinoplasty? J Oral Maxillofac Surg. 2005 Aug;63(8):1088-90. doi: 10.1016/j.joms.2005.04.008. PMID 16094573